CLINICAL TRIAL: NCT01285505
Title: Open-Label, Randomized, Single-Dose, 2-Way Crossover Bioequivalence Study Comparing A New Alprazolam Sublingual Tablet Formulation To An Alprazolam Sublingual Tablet
Brief Title: Bioequivalence of a New and a Commercial Alprazolam Sublingual Formulation
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A6131020
Record Dates: First submitted 2011-01-26; First posted 2011-01-28 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: alprazolam; sublingual; bioequivalence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alprazolam commercial sublingual tablet (Active Comparator)
  Interventions: Drug: alprazolam commercial sublingual formulation
- Alprazolam test sublingual tablet (Experimental)
  Interventions: Drug: alprazolam test sublingual tablet

INTERVENTIONS:
Drug: alprazolam commercial sublingual formulation — 0.5 mg tablet, single dose
  Arms: Alprazolam commercial sublingual tablet
Drug: alprazolam test sublingual tablet — 0.5 mg tablet, single dose
  Arms: Alprazolam test sublingual tablet

SUMMARY:
This study tests the hypothesis that the bioavailability of alprazolam from a new sublingual formulation is the same as that from an existing sublingual formulation.

ELIGIBILITY:
Inclusion Criteria:

* healthy male or female subjects
* BMI 18 to 26.9
* must give informed consent

Exclusion Criteria:

* clinically significant disease
* narrow angle glaucoma
* positive drug screen

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Alprazolam bioavailability as assessed from the area under the concentration-time curve (AUC) | 11 days
Alprazolam bioavailability as assessed by peak concentration (Cmax) | 11 days

SECONDARY OUTCOMES:
Alprazolam time of maximum concentration (Tmax) | 11 days
Half life of alprazolam | 11 days
Clinically significant safety laboratory tests | 11 days
Clinically significant adverse events | 11 days
Clinically significant vital signs | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6131020&StudyName=Bioequivalence%20of%20a%20new%20and%20a%20commercial%20alprazolam%20sublingual%20formulation